CLINICAL TRIAL: NCT07259837
Title: Association Between Preoperative Health and Functional Status and Postoperative Complications in Elderly Patients: An Analysis of a Prospective Cohort
Brief Title: Association Between Preoperative Health and Functional Status and Postoperative Complications in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yanhong Liu, Deputy Chief of administration, Anesthesiology, Chinese PLA General Hospital
Other Study IDs: PLAGH - SCALE
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Functional Status; Postoperative Complications; Older Adults (65 Years and Older)
Keywords: Functional status; Quality of life; Major Adverse Cardiac and Cerebrovascular Events; Older adults
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A retrospective cohort study based on prospectively collected data.: Patients were divided into the MACCE group and the non-MACCE group according to the occurrence of major adverse cardiac and cerebrovascular events within 30 days after surgery.

SUMMARY:
Using prospectively collected clinical data from the Chinese Perioperative Database of Elderly Patients, this study retrospectively analyzed patients aged ≥65 years who underwent elective non-cardiac, non-neurosurgical procedures under general anesthesia between April 2020 and April 2022. The study examined the associations between various preoperative health and functional status assessment tools and the occurrence of cardiovascular and cerebrovascular complications within 30 days after surgery, aiming to compare the clinical value of different assessment instruments.

ELIGIBILITY:
Inclusion criteria:

1. Aged ≥65 years;
2. Scheduled for elective non-cardiac, non-neurosurgical procedures;
3. Consented to undergo preoperative functional status and quality of life assessments.

Exclusion criteria:

1. Had severe dementia, language disorders, significant hearing or visual impairments, or were in a coma;
2. Had Mini-Mental State Examination (MMSE) scores below the established educational thresholds: <18 for illiterate individuals, <21 for those with primary education (≤6 years), and <25 for those with secondary education or higher (>6 years);
3. Underwent local anesthesia or monitored anesthesia care;
4. Had an operative time ≤30 minutes;
5. Incompleted all the designated functional status and quality of life assessments.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients were interviewed one day before surgery and completed a comprehensive preoperative functional status and quality of life assessment, which included the Basic Activities of Daily Living (BADL), Instrumental Activities of Daily Living (IADL), EuroQol Five-Dimension Five-Level (EQ-5D-5L), Metabolic Equivalent of Task (MET), and FRAIL scale.
Sampling Method: Non-Probability Sample
Enrollment: 8751 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the occurrence of MACCE within 30 days after surgery. | Within 30 days after surgery.
  The primary outcome was the occurrence of MACCE within 30 days after surgery, defined as any of the following: stroke, myocardial infarction, angina pectoris, congestive heart failure, cardiac arrest, or all-cause mortality.[33] Postoperative complications were systematically assessed on days 1-5, 7, and 30, and continued until discharge. For discharged patients, outcomes were recorded via telephone follow-up, with diagnoses from the treating hospital. For MACCE, postoperative medical records of hospitalized patients were thoroughly reviewed according to the follow-up schedule, including serial measurements of serum myocardial injury biomarkers, electrocardiograms, echocardiograms, coronary angiography findings, postoperative progress notes, consultation records, and expert diagnostic evaluations.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided